CLINICAL TRIAL: NCT06373926
Title: Evaluation of Cell Membrane Expression of Annexin A2 on Monocytes by Flow Cytometry in Primary Antiphospholipid Syndrome
Acronym: MONOCYTAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2019_843_0010
Record Dates: First submitted 2024-04-09; First posted 2024-04-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Antiphospholipid Syndrome
Keywords: annexin A2; antiphospholipid syndrome; monocytes
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Experimental): APS patients
  Interventions: Biological: blood withdrawal
- control (Active Comparator): healthy individuals
  Interventions: Biological: blood withdrawal

INTERVENTIONS:
Biological: blood withdrawal — blood withdrawal

SUMMARY:
Annexin A2 (ANXA2), an endothelial cell receptor for plasminogen and tissue plasminogen activator, plays a pivotal role in regulation of fibrinolysis in vitro and in vivo and has been identified as a new autoantigen in antiphospholipid syndrome (APS). ANXA2 can exist as a monomer or a heterotetrameric complex with S100A10 protein. The aim of this study was to evaluate the cell membrane expression of ANXA2 on circulating monocytes in APS by flow cytometry. Several pathogenic mechanisms are involved in APS such as activation of endothelial cells, platelets and monocytes, inhibition of the natural anticoagulant protein C/protein S pathway, activation of the complement system and also impairment of fibrinolysis. Annexin A2 which hits binding partner S100A10, ANXA2 forms a cell surface complex that regulates generation of plasmin. ANXA2 is involved in the pathogenesis of APS-associated through several possible mechanisms. Human peripheral blood monocytes represent the major circulating ANXA2-expressing cell and ANXA2-mediated assembly of plasminogen and tissue activator of plasminogen (tPA) on monocyte/macrophages contributes to plasmin generation. Thus the investigators could suppose that decrease of cell membrane expression of ANXA2 on circulating monocytes represent a new pathogenic mechanism in APS.

ELIGIBILITY:
Inclusion Criteria:

* APS patients who fulfilled the revised criteria for APS

Exclusion Criteria:

* Patients less than 18 years old
* Solid and hematological malignancies
* Other autoimmune diseases
* Cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Cell membrane expression rate of ANXA2 on circulating monocytes in APS | 1 hour

SECONDARY OUTCOMES:
Cellular expression of ANXA2 and S100A10 in APS patients | 1 hour
cell membrane expression of ANXA2 and S100A10 in APS patients | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No